CLINICAL TRIAL: NCT02596568
Title: The Use of Transcranial Direct Current Stimulation During Slow Wave Sleep in Healthy Students and Older Adults
Brief Title: The Effect of tDCS Applied During Sleep on Memory Consolidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00020393
Record Dates: First submitted 2014-03-13; First posted 2015-11-04 (Estimated); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Sleep
MeSH Terms: interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS stimulation (Experimental): Anodal tDCS will be applied bi-frontally using Chattanooga Ionto™ Iontophoresis System - Phoresor. A square wave will be delivered at 0.75 Hz for five blocks of five minutes each with one minute inter-train interval. Stimulation will be applied following 8 epochs of consecutive stage 2 or deeper sleep.
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Sham tDCS stimulation (Sham Comparator): tDCS electrodes will be applied bi-frontally using Chattanooga Ionto™ Iontophoresis System - Phoresor, however stimulation will never be turned on.
  Interventions: Other: Sham

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS is a type of brain stimulation that uses low current applied directly over the scalp to increase, or decrease cortical activity under the stimulating electrodes. tDCS applied bi-frontally using Chattanooga Ionto™ Iontophoresis System - Phoresor. A square wave will be delivered at 0.75 Hz for five blocks of five minutes each with one minute inter-train interval. Stimulation will be applied following 8 epochs of consecutive stage 2 or deeper sleep.
  Arms: Active tDCS stimulation
Other: Sham — tDCS device connected and tested, but not turned on during the night. This has been found to be an effective sham in other studies using this technique.
  Arms: Sham tDCS stimulation

SUMMARY:
This study will attempt to use a type of non-invasive brain stimulation technology during sleep to improve measures of sleep quality and memory in young healthy students and older adults. The type of brain stimulation is called transcranial direct current stimulation (tDCS), which uses small currents of electricity to increase or decrease the activity of specific areas of the brain.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a safe, non-invasive, and inexpensive brain stimulation modality that has been shown to have the ability to modulate both cortical and deep brain structure activity. This technique has undergone a significant amount of investigation in varied neuropsychiatric populations and interest in this technique has increased dramatically as of late.

Some researchers have studied the effects of this modality on sleep as well as memory with promising results. One such study demonstrated that by using bilateral tDCS with a pattern of stimulation in the delta frequency range (0-3 Hz) delivered during slow wave sleep, that it is possible to increase delta power during slow wave sleep, as well as improve sleep efficiency. In addition to showing that it is possible to enhance slow waves, it was also demonstrated that this increase was associated with an improvement of a measure of declarative memory consolidation (one of the theorized functions of slow wave sleep). Enhancing memory function in a normal healthy group raises the possibility that it would also be possible to enhance memory in clinical populations who would benefit from such an intervention.

The investigators propose to test this intervention for replication in a similar cohort.

ELIGIBILITY:
Inclusion Criteria:

* Students
* Adults aged 60 or greater.

Exclusion Criteria:

* If they are taking any prescription or over the counter medications.
* If they have any currently active neurologic, psychiatric, hormonal, metabolic, circulatory, or sleep disturbances. -They must specifically not have a history of seizures, closed head injuries with loss of consciousness for greater than 5 minutes, any known brain tumors or lesions, metal implants or implanted devices above the neck, a history of eczema, or other sensitive conditions, or an allergy to latex.
* They must not smoke cigarettes, use illicit drugs, or meet criteria for alcohol abuse or dependence in their lifetime defined by SCID criteria.
* They must be free of alcohol for at least 48 hours prior to each night of the study
* They must not consume more than the equivalent of 500mg of caffeine daily.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Declarative memory assessed by paired word association test | Pre sleep/intervention, and post sleep/intervention
  Prior to and directly after a night of sleep we will assess declarative memory using a paired word association tests. In the pre-sleep assessment there will be a learning phase where the word list will be presented serially, until 60% of the words are retained. In the post sleep assessment the word list will be given again once. The outcome measure is the change in words retained between pre and post sleep assessments. Subsequently the followup interval is approximately 8-9 hours with baseline before bedtime, and follow up assessment once the patient is awoken.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sahlem, M.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States